CLINICAL TRIAL: NCT00486512
Title: A Clinical Trial Evaluating the Efficacy and Safety of a Combination Treatment Administered Over 3 Years in Patients at Risk of Experiencing Recurrence of Colorectal Adenomas
Brief Title: Chemoprevention of Colorectal Adenomas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall program was terminated
Sponsor: Colotech A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COLO CP-01-US
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Adenomatous Polyps
Keywords: colorectal, adenomas, prevention
MeSH Terms: conditions — Adenomatous Polyps; Adenoma | interventions — Calcitriol; Aspirin; Calcium Carbonate; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (calcitriol+ASA+CaCO3) (Experimental): Daily dose of 0.5 mg calcitriol (1a -25-dihydroxycholecalciferol, Rocaltrol; Roche, Basel, Switzerland), 75 mg acetylsalicylic acid (ASA), and 1250 mg calcium carbonate (CaCO3). The daily dose was administered as 1 capsule containing 0.5 mg calcitriol (Rocaltrol; Roche) and 2 tablets containing a 37.5-mg ASA core with a 625-mg calcium carbonate shell (tablet-in-tablet) that was made expressly for this study. Patients should take 1 capsule and 2 tablets daily, together or separately. Timing of the intake is not important; study medication can be taken with or without food. The daily dose should not be exceeded. Before randomization, patients were given the placebo and followed up for a 3-week run-in period. Only patients who showed a placebo medication compliance rate of at least 80% were eligible for randomization. The primary outcome was the proportion of patients with recurrence of any adenomas as detected by colonoscopy after 3 years of treatment.
  Interventions: Drug: 0.5 mg calcitriol (1a -25-dihydroxycholecalciferol); Drug: 75 mg acetylsalicylic acid (ASA) + 1250 mg calcium carbonate (CaCO3); Procedure: Colonoscopy
- Placebo to calcitriol+ASA+CaCO3 (Placebo Comparator): Daily dose of matching placebo to 0.5 mg calcitriol, 75 mg acetylsalicylic acid (ASA), and 1250 mg calcium carbonate (CaCO3). Patients should take 1 capsule and 2 tablets of placebo daily, together or separately. Timing of the intake is not important; study medication can be taken with or without food. The daily dose should not be exceeded. Before randomization, patients were given the placebo and followed up for a 3-week run-in period. Only patients who showed a placebo medication compliance rate of at least 80% were eligible for randomization. The primary outcome was the proportion of patients with recurrence of any adenomas as detected by colonoscopy after 3 years of treatment.
  Interventions: Drug: placebo to 0.5 mg calcitriol (1a -25-dihydroxycholecalciferol); Drug: placebo to 75 mg acetylsalicylic acid (ASA) + 1250 mg calcium carbonate (CaCO3); Procedure: Colonoscopy

INTERVENTIONS:
Drug: 0.5 mg calcitriol (1a -25-dihydroxycholecalciferol)
  Arms: Active Treatment (calcitriol+ASA+CaCO3)
Drug: 75 mg acetylsalicylic acid (ASA) + 1250 mg calcium carbonate (CaCO3)
  Arms: Active Treatment (calcitriol+ASA+CaCO3)
Drug: placebo to 0.5 mg calcitriol (1a -25-dihydroxycholecalciferol)
  Arms: Placebo to calcitriol+ASA+CaCO3
Drug: placebo to 75 mg acetylsalicylic acid (ASA) + 1250 mg calcium carbonate (CaCO3)
  Arms: Placebo to calcitriol+ASA+CaCO3
Procedure: Colonoscopy

SUMMARY:
The purpose of the study is to investigate if long-term treatment with three known drugs (acetylsalicylic acid, 1α 25-dihydroxy cholecalciferol, and calcium carbonate) prevents recurrence of colorectal adenomas.

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel group, prospective, double blind, placebo controlled clinical trial of chemoprevention in patients at increased risk of developing colorectal cancer (CRC). The Colotech combination treatment (acetylsalicylic acid, 1α 25-dihydroxy cholecalciferol, and calcium carbonate) will be compared to placebo with regards to safety and efficacy during 3 years of treatment. The randomized treatment period will be preceded by a 3-week single blind placebo run-in period, which will assess patient's compliance to treatment. In order to collect data on the durability of treatment effect, follow-up data from a surveillance colonoscopy will be collected two years after the 3-year colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 40-75 years of age, both sexes.
* Colonoscopy including the cecum at trial entry
* The removed adenoma(s) have be to tubular, tubulovillous or villous, and fulfill one of the three following criteria:

  1. one adenoma with diameter ≥ 1 cm
  2. ≥ 2 adenomas of any size
  3. an adenoma of any size and familial disposition for colorectal cancer, as long as the person is a first degree relative with a colorectal cancer patient

Exclusion Criteria:

* Familial Adenomatous Polyposis Syndrome
* Member of a family with hereditary non-polyposis colorectal cancer (HNPCC)
* Proctocolectomy (colonic and/or rectum resection permitted).
* Inflammatory bowel disease (Crohn´s disease, Ulcerative Colitis).
* Ischemic cardiovascular disease.
* Patients with known gastro-duodenal ulcer at time of inclusion.
* Cancer within the past 5 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2007-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assessment of cumulative frequency of recurrence of colorectal adenomas post ablation | 156 weeks
  The purpose of the study is to investigate if long-term treatment with three known drugs (acetylsalicylic acid, 1α 25-dihydroxy cholecalciferol, and calcium carbonate) prevents recurrence of colorectal adenomas which were removed during colonoscopy.

SECONDARY OUTCOMES:
Assessment of number and size of colorectal adenomas measured after three years of chemoprevention using the study drug | 3 years
  The purpose of the study is to investigate if long-term treatment with three known drugs (acetylsalicylic acid, 1α 25-dihydroxy cholecalciferol, and calcium carbonate) prevents recurrence of colorectal adenomas which were removed during colonoscopy.
Assessment of durability of polyp-free colon post surgical ablation for two years post-treatment with chemoprevention with study drug | additional 2 years
  The purpose of the study is to investigate if long-term treatment with three known drugs (acetylsalicylic acid, 1α 25-dihydroxy cholecalciferol, and calcium carbonate) prevents recurrence of colorectal adenomas which were removed during colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Raskov, M.D., Study Director — Colotech A/S
Locations (39):
- United States (24):
  - Alabama Digestive Disorders Center, P.C., Huntsville, Alabama
  - San Diego Digestive Disease Consultants, Inc., San Diego, California
  - Advance Digestive Care, Clearwater, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Atlanta Center for Gastroenterology, PC, Decatur, Georgia
  - Central Indiana Gastroenterology Group, Anderson, Indiana
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Gastroenterology Associates of Eastern Maine, Bangor, Maine
  - Digestive Disorders Associates, Annapolis, Maryland
  - Office of Alan A. Rosen, M.D., Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Colon and Rectal Surgery Associates, Ltd., Saint Paul, Minnesota
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Gastroenterology Research Associates, Cedar Knolls, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Digestive Health Specialists PA, Winston-Salem, North Carolina
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - Regional Gastroenterology Associates of Lancaster, Ltd, Lancaster, Pennsylvania
  - North Texas Gastroenterology Consultants, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Advanced Healthcare, S.C., Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Russia (15):
  - Russian Center of Functional Surgical Gastroenterology, Krasnodar
  - Federal State Enterprise "Russian Federation Defense Ministry Burdenko Main Military Clinical Hospital", Moscow
  - Out-patient clinic No. 2 of the Administration for the President of Russian Federation, Moscow
  - State Medical Stomatological University, Moscow
  - Out-patient clinic No. 3 of the Administration for the President of Russian Federation, Moscow
  - Rostov State Medical University, Rostov-on-Don
  - 2nd Terapy Department Military Medical Academy, Saint Petersburg
  - All Russian Center of Emergency and Radiation Medicine of EMERCOM of Russia, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - St. Petersburg Central Medical Sanitary Department of Federal Biological Agency, Saint Petersburg
  - Saint-Petersburg State City Hospital No 26, Saint Petersburg
  - Dept of Gastroenterology and Nutrition, Saint Petersburg
  - Smolensk City Clinical Hospital No 1, Smolensk
  - Stavropol State Medical Academy, Stavropol
  - Yaroslav City Clinical Hospital No 2, Yaroslavl

REFERENCES:
- [Derived] Pommergaard HC, Burcharth J, Rosenberg J, Raskov H. Aspirin, Calcitriol, and Calcium Do Not Prevent Adenoma Recurrence in a Randomized Controlled Trial. Gastroenterology. 2016 Jan;150(1):114-122.e4. doi: 10.1053/j.gastro.2015.09.010. Epub 2015 Sep 25. PMID 26404953
- [Derived] Carroll C, Cooper K, Papaioannou D, Hind D, Pilgrim H, Tappenden P. Supplemental calcium in the chemoprevention of colorectal cancer: a systematic review and meta-analysis. Clin Ther. 2010 May;32(5):789-803. doi: 10.1016/j.clinthera.2010.04.024. PMID 20685491